CLINICAL TRIAL: NCT00185341
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Safety, Tolerability and Efficacy of the CCR1 Antagonist ZK 811752, Given Orally in a Dose of 600 mg Three Times Daily, for the Treatment of Endometriosis Over 12 Weeks
Brief Title: Study to Investigate the Efficacy of a Non-hormonal Drug Against Endometriosis Associated Pelvic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91399; 2004-000630-37 (EudraCT Number); 308601
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Endometriosis
Keywords: Endometriosis associated pelvic pain
MeSH Terms: conditions — Endometriosis | interventions — BX 471

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- CCR-1 Receptor Antagonist (Experimental): Subjects received 600 mg (2 x 300 mg tablets) of CCR-1 Receptor Antagonist 3 times daily
  Interventions: Drug: CCR1-Antagonist (BAY86-5047, ZK811752)
- Placebo (Placebo Comparator): Subjects received placebo corresponding to verum
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CCR1-Antagonist (BAY86-5047, ZK811752) — Given orally in a dose of 600 mg three times daily over 12 weeks
  Arms: CCR-1 Receptor Antagonist
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study was designed as a proof-of-concept trial to evaluate safety, tolerability, and the efficacy of 1800 mg (ZK 811752 600 mg given orally three times daily) over 12 weeks for the treatment of endometriosis associated pelvic pain (EAPP) in comparison to placebo.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Pain associated with proven endometriosis, as determined by diagnostic measures within 24 months prior to start of treatment
* Women with cyclic menstrual bleeding- Good general health
* Willingness to use a barrier contraceptive method such as condoms but no hormonal contraception- Willingness to use only up to 3 Ibuprofen 400 tablets as pain killer for endometriosis-related pelvic pain - Age 18 to 45 years inclusive - Fertile and non-fertile Exclusion Criteria:
* Pregnancy, lactation- Bearing of an intra-uterine device
* Current use of hormonal agents.
* Actual or history of cardiovascular and further serious disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2005-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Individual absolute change in endometriosis associated pelvic pain (EAPP) | 12 weeks
  EAPP was assessed by a composite parameter, consisting of the reading of the visual analog scale (VAS) and the intake of rescue medication
Individual change in intake of rescue medication | 12 weeks

SECONDARY OUTCOMES:
Number of participants with adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (27):
- Czechia (2):
  - Hradec Králové
  - Prague
- Denmark (2):
  - Aarhus
  - Glostrup Municipality
- Finland (5):
  - Helsinki
  - Joensuu
  - Kuopio
  - Oulu
  - Turku
- France (3):
  - Bordeaux, France
  - Clermont-Ferrand
  - Lyon
- Netherlands (3):
  - Amsterdam
  - Maastricht
  - Nijmegen
- Spain (6):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Oviedo, Principality of Asturias
  - Valencia, Valencia
  - Barcelona
  - Seville
- Sweden (6):
  - Stockholm, Sweden
  - Gothenburg
  - Lund
  - Skövde
  - Stockholm
  - Uppsala

REFERENCES:
- [Derived] Sieverding M, Gerlinger C, Seitz C. Substituting a randomised placebo control group with a historical placebo control in an endometriosis pain trial: a case study re-evaluating trial data using historical control data from another trial. BMJ Open. 2023 Jul 21;13(7):e063188. doi: 10.1136/bmjopen-2022-063188. PMID 37479520
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/